CLINICAL TRIAL: NCT03897855
Title: Memory Inhibition and Delayed Onset Post-traumatic Stress Disorder in Older Subjects
Acronym: I-TSPT-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Niort (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CH-NIORT-2018-02
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Post-Traumatic Stress Disorder in Old Age

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (TSPT-R) (Other): Post Traumatic Stress Disorder
  Interventions: Other: Post Traumatic Stress Disorder
- control (Experimental): No Post Traumatic Stress Disorder
  Interventions: Other: Post Traumatic Stress Disorder

INTERVENTIONS:
Other: Post Traumatic Stress Disorder — The test "Think / No-Think"

SUMMARY:
In the elderly, we can see a post-traumatic syndrome associated with an event that occurred before old age that had not previously manifested or not fully manifested.

This little-known pathology and notable psychiatric co-morbidities (depression, anxiety) can take in elderly subjects different masks that interfere with diagnosis and treatment.

The data in the literature suggest that this Post-Traumatic Stress Disorder with Delayed Expression (TSPT-R) may be related to a deficiency of the executive functions of inhibition, and more particularly a deficit of mental memory inhibition and therefore the removal of unwanted memories.

ELIGIBILITY:
Inclusion Criteria:

-

Regarding the constitution of the group patient (TSPT-R):

* Subjects 65 years of age or older
* Clinical diagnosis of delayed-onset PTSD according to DSM-5 criteria after 65 years
* The traumatic event must have taken place at the latest before 65 years
* Affiliated person or beneficiary of a social security scheme.
* Written consent before any examination required by research)

Regarding the constitution of the control group:

* Subjects 65 years of age or older
* No diagnosis of PTSD (delayed or not) or history of PTSD (delayed or not)
* Affiliated person or beneficiary of a social security scheme.
* Written consent before any examination required by the research).

Exclusion Criteria:

* For both groups:
* Acute or chronic cognitive impairment known
* GRECO MMSE pathological score less than or equal to the pathological threshold weighted according to level of education and age, namely:

  * 22 if no diploma
  * 23 if certificate of study
  * 25 if patent
  * 26 if bin or more
  * Remove one point at each threshold if age> 80 years
* Sensory or motor disorder preventing the passing of different tests
* Psychotic disorder
* Mood disorder in decompensation (for depression, HAD-D score equal to or greater than 11)
* Disorder of the use of a moderate or severe substance (except tobacco).
* Patients under guardianship or curatorship.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Inhibition score measured by the Think / No-Think Test | 1 month
  the average of the inhibition score measured by the "Think / No-Think" test as defined by Anderson and Green (2001) and then reviewed by Anderson et al. in 2011

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LEGER, Doctor, Study Director — Centre Hospitalier de Niort
Locations (1):
- Centre Hospitalier de Niort, Niort, France